CLINICAL TRIAL: NCT02139696
Title: Does Targeting of Sphingosine-1 Phosphate Receptors Reduce Microglial Activation in Multiple Sclerosis? A [11C]PK11195 Brain PET Study
Brief Title: Sphingosine-1 Phosphate -Receptor Targeting and Microglial Activation
Acronym: FINGOPET
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FINGOPET
Record Dates: First submitted 2014-05-08; First posted 2014-05-15 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MS patients initiating fingolimod: Patients will be imaged using PET and MRI at baseline, and twice during treatment.
  Interventions: Radiation: PET and MRI

INTERVENTIONS:
Radiation: PET and MRI — Patients will be imaged using PET and MRI at baseline, and twice during treatment

SUMMARY:
To evaluate the usability of positron emission tomography imaging as a novel outcome measure in multiple sclerosis studies

DETAILED DESCRIPTION:
Background and Rationale

In multiple sclerosis (MS), significant pathology correlating to disease progression, to expanded disability status scale (EDSS) and to cognitive decline, takes place outside the plaque areas, i.e. in areas of normal appearing white matter and gray matter. Neuropathological studies suggest that mechanisms involved in this widespread pathology include activation of microglial cells, oxidative stress and deficiency in mitochondrial functions. Activated microglia can be detected in vivo with a translocator protein (TSPO), expressed in activated, but not resting microglia) binding radioligands and positron emission tomography (PET). 11Carbon-PK11195 radioligand is one such radioligand. Importantly, the possible effect of MS therapies on microglial activity can be evaluated in patients in vivo with PET-imaging performed before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

Having signed the informed consent of the investigator-initiated PET study

* Age 18 - 58 years at the time of informed consent.
* MS according to Poser or McDonald criteria
* EDSS score from 0.0 to 6.5.
* Moderate to heavy lesion load ( >9 T2 lesions) in MRI

Exclusion Criteria:

* - Patients with other neurodegenerative disease than MS
* Disease modifying therapy (DMT) within 4 weeks of imaging
* Corticosteroid treatment within 4 weeks of imaging
* Patients with significant abnormal findings other than MS in the screening MRI.
* Patients with claustrophobia, or a history of moderate to severe anxiety disorder or panic attacks (which could potentially lead to preterm termination of the imaging)
* Contraindication to PET scan investigations
* Exposure to experimental radiation in the past 12 months such that radiodosimetry limits would be exceeded by participating in this study.
* Intolerance to previous PET scans; i.e. previous hypersensitivity reactions to any PET ligand or imaging agent or failure to participate in and comply with previous PET scans.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 10 patients with multiple sclerosis who will be initiated on fingolimod in the neurology outpatient clinic of the Turku University hospital in Turku, Finland.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change of 11C-PK11195-radioligand binding using PET | 0 to 24 weeks
  Patients will be switched to fingolimod from first-line therapies as per indication and as part of their normal treatment regimen, and those who will consent to participate in this investigator-initiated PET study, will be imaged at baseline (pre-treatment phase) and after 6-8 weeks and 24 weeks of treatment. Purpose is to compare the binding of the radioligand between these three time points.

SECONDARY OUTCOMES:
MRI metrics | 0, 6-8 wk, 24 wk
  To evaluate the total lesion load of the white matter MS plaques with MRI; baseline vs. 6-8 weeks vs. 24 weeks of Gilenya treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laura Airas, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rissanen E, Tuisku J, Rokka J, Paavilainen T, Parkkola R, Rinne JO, Airas L. In Vivo Detection of Diffuse Inflammation in Secondary Progressive Multiple Sclerosis Using PET Imaging and the Radioligand (1)(1)C-PK11195. J Nucl Med. 2014 Jun;55(6):939-44. doi: 10.2967/jnumed.113.131698. Epub 2014 Apr 7. PMID 24711650